CLINICAL TRIAL: NCT00842296
Title: ClosureFAST - Endovascular Radiofrequency Great Saphenous Vein Treatment Using a Catheter With an Integrated Heating Element
Brief Title: ClosureFAST - Radiofrequency Great Saphenous Vein Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Endovascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLF-05-03
Record Dates: First submitted 2009-02-10; First posted 2009-02-12 (Estimated); Results first posted 2017-12-11 (Actual); Last update posted 2018-03-12 (Actual); Status verified 2018-02

CONDITIONS: Venous Reflux
Keywords: GSV; RadioFrequency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Seg. RF Ablation with CLF catheter (Experimental): Single Arm with CLF Catheter
  Interventions: Device: RF ablation (ClosureFAST)

INTERVENTIONS:
Device: RF ablation (ClosureFAST) — Segmental RF Ablation with the CLF catheter
  Other Names: CLF; CLosureFAST

SUMMARY:
The purpose of this study is to confirm that the ClosureFAST system can be used as an alternative to the current ClosurePlus catheter for treating the GSV and to accumulate pivotal data for optimization of the operating parameters.

DETAILED DESCRIPTION:
The purpose of this study is to confirm that the ClosureFAST system can be used as an alternative to the current ClosurePlus catheter for treating the GSV and to accumulate pivotal data for optimization of the operating parameters. The results from this study will be used to further evaluate the risks and benefits of the ClosureFAST device and to obtain clinical evidence that the treatment provides effective and durable clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years of age at the time of enrollment
* Symptomatic lower limb venous disease involving the GSV

Exclusion Criteria:

* Thrombosis in the vein segment to be treated
* Known or suspected pregnancy or actively breast feeding at time of treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 326 (Actual)
Dates: Start 2006-04; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Hasenbank, PhD, Study Director — Medtronic

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Proebstle TM, Mohler T. A longitudinal single-center cohort study on the prevalence and risk of accessory saphenous vein reflux after radiofrequency segmental thermal ablation of great saphenous veins. J Vasc Surg Venous Lymphat Disord. 2015 Jul;3(3):265-9. doi: 10.1016/j.jvsv.2014.10.001. Epub 2014 Dec 6. PMID 26992304

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment from April 24, 2006- September 5, 2006. Medical offices/clinics and university hospital.
Units Other Than Participants: limbs
Groups:
- ClosureFAST® - Endovascular Radiofrequency Great Saphenous Vei: Single Arm with ClosureFAST (CLF) Catheter with an integrated healing element. Radiofrequency (RF) ablation (ClosureFAST): Segmental RF Ablation with the CLF catheter
Period: Overall Study
Arm/Group | ClosureFAST® - Endovascular Radiofrequency Great Saphenous Vei
Started | 326; 396 limbs
Completed | 326; 396 limbs
Not Completed | 0; 0 limbs

BASELINE CHARACTERISTICS:
Population: 326 patients were enrolled and 396 limbs were treated and are analyzed. Only 395 limbs provided baseline CEAP data.
Units Other Than Participants: limbs
Arm/Group | ClosureFAST® - Endovascular Radiofrequency Great Saphenous Vei
Number analyzed (Participants) | 326
Number analyzed (limbs) | 396
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.8 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 239
  Male | 87
Region of Enrollment [Number; unit: participants]
  United States | 101
  Europe | 225
CEAP [Number; unit: limbs] — CEAP (Clinical/Etiology/Anatomy/Pathophysiology) Clinical Score:
  C0: No visible/palpable sign C1: Reticular spider veins C2: Simple varicose veins C3: Ankle edema C4: Skin pigmentation C5: Healed venous ulcer C6: Open venous ulcer
  395 out of 396 limbs reported a Baseline CEAP score. Population: only 395 out of 396 limbs reported a Baseline CEAP score
  limbs
    number analyzed (limbs) | 395
    C0 | 1
    C1 | 5
    C2 | 213
    C3 | 110
    C4 | 60
    C5 | 4
    C6 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Limbs Without Vein Occlusion
Description: Defined as the absence of flow in the treated vein as documented on the post-procedure and follow-up Duplex Ultrasound (DU) scan. Flow which originates in the Saphenofemoral Junction (SFJ) and which measures < 3 cm in length, does not constitute a failure.
Time Frame: 6 Months
Population: 363 limbs were available for primary outcome measure evaluation at the 6M timepoint.
Measure: Mean (Standard Error); unit: percentage of limbs
Units Other Than Participants: limbs
Arm/Group | ClosureFAST® - Endovascular Radiofrequency Great Saphenous Vei
Number analyzed (Participants) | 293
Number analyzed (limbs) | 363
percentage of limbs | 97.6 (0.8)

2. Primary Outcome: Percentage of Limbs Without Vein Occlusion
Description: Defined as the absence of flow in the treated vein as documented on the post-procedure and follow-up DU scan. Flow which originates in the SFJ and which measures < 3 cm in length, does not constitute a failure.
Time Frame: 12 months
Population: 350 limbs were evaluated at the 12M timepoint
Measure: Mean (Standard Error); unit: percentage of limbs
Units Other Than Participants: limbs
Arm/Group | ClosureFAST® - Endovascular Radiofrequency Great Saphenous Vei
Number analyzed (Participants) | 280
Number analyzed (limbs) | 350
percentage of limbs | 96.6 (0.9)

3. Primary Outcome: Percentage of Limbs Without Vein Occlusion
Description: Vein occlusion is defined as the absence of flow in the treated vein as documented on the post-procedure and each successive follow-up DU scan.
Time Frame: 2 years
Population: Out of the limbs treated 329 limbs were available for a Duplex Ultrasound scan at the 2Y follow-up
Measure: Mean (Standard Error); unit: percentage of limbs
Units Other Than Participants: limbs
Arm/Group | ClosureFAST® - Endovascular Radiofrequency Great Saphenous Vei
Number analyzed (Participants) | 263
Number analyzed (limbs) | 329
percentage of limbs | 94.3 (1.2)

4. Primary Outcome: Percentage of Limbs Without Vein Occlusion
Description: as for outcome 2
Time Frame: 3 years
Population: 293 limbs were evaluated at the 3Y timepoint
Measure: Mean (Standard Error); unit: percentage of limbs
Units Other Than Participants: limbs
Arm/Group | ClosureFAST® - Endovascular Radiofrequency Great Saphenous Vei
Number analyzed (Participants) | 229
Number analyzed (limbs) | 293
percentage of limbs | 92.8 (1.4)

5. Primary Outcome: Percentage of Limbs Without Vein Occlusion
Description: as for outcome 2
Time Frame: 4 years
Population: 275 limbs were evaluated at the 4Y timepoint
Measure: Mean (Standard Error); unit: Percentage of limbs
Units Other Than Participants: limbs
Arm/Group | ClosureFAST® - Endovascular Radiofrequency Great Saphenous Vei
Number analyzed (Participants) | 210
Number analyzed (limbs) | 275
Percentage of limbs | 91.1 (1.5)

6. Primary Outcome: Percentage of Limbs Without Vein Occlusion
Description: as for outcome 2
Time Frame: 5 years
Population: 279 limbs were evaluated at the 5Y timepoint
Measure: Mean (Standard Error); unit: Percentage of limbs
Units Other Than Participants: limbs
Arm/Group | ClosureFAST® - Endovascular Radiofrequency Great Saphenous Vei
Number analyzed (Participants) | 221
Number analyzed (limbs) | 279
Percentage of limbs | 90.0 (1.7)

7. Primary Outcome: Percentage of Limbs Without Reflux in the Treated Vein Segment
Description: No reflux in the vein segment treated. Reflux was defined as reversal flow >0.5s with subject standing or in reverse Trendelenburg position of at least 15° after distal augmentation.
Time Frame: 6 months
Population: 363 limbs were evaluated at the 6M timepoint
Measure: Mean (Standard Error); unit: Percentage of limbs
Units Other Than Participants: limbs
Arm/Group | ClosureFAST® - Endovascular Radiofrequency Great Saphenous Vei
Number analyzed (Participants) | 293
Number analyzed (limbs) | 363
Percentage of limbs | 99.5 (0.4)

8. Primary Outcome: Percentage of Limbs Without Reflux in the Treated Vein Segment
Description: as for outcome 7
Time Frame: 12 months
Population: 350 limbs were evaluated at the 12M timepoint
Measure: Mean (Standard Error); unit: Percentage of limbs
Units Other Than Participants: limbs
Arm/Group | ClosureFAST® - Endovascular Radiofrequency Great Saphenous Vei
Number analyzed (Participants) | 280
Number analyzed (limbs) | 350
Percentage of limbs | 98.9 (0.5)

9. Primary Outcome: Percentage of Limbs Without Reflux in the Treated Vein Segment
Description: as for outcome 7
Time Frame: 2 years
Population: 329 limbs were evaluated at the 2Y timepoint
Measure: Mean (Standard Error); unit: Percentage of limbs
Units Other Than Participants: limbs
Arm/Group | ClosureFAST® - Endovascular Radiofrequency Great Saphenous Vei
Number analyzed (Participants) | 263
Number analyzed (limbs) | 329
Percentage of limbs | 97.8 (0.8)

10. Primary Outcome: Percentage of Limbs Without Reflux in the Treated Vein Segment
Description: as for outcome 7
Time Frame: 3 years
Population: 293 limbs were evaluated at the 3Y timepoint
Measure: Mean (Standard Error); unit: Percentage of limbs
Units Other Than Participants: limbs
Arm/Group | ClosureFAST® - Endovascular Radiofrequency Great Saphenous Vei
Number analyzed (Participants) | 229
Number analyzed (limbs) | 293
Percentage of limbs | 95.7 (1.1)

11. Primary Outcome: Percentage of Limbs Without Reflux in the Treated Vein Segment
Description: as for outcome 7
Time Frame: 4 years
Population: 275 limbs were evaluated at the 4Y timepoint
Measure: Mean (Standard Error); unit: Percentage of limbs
Units Other Than Participants: limbs
Arm/Group | ClosureFAST® - Endovascular Radiofrequency Great Saphenous Vei
Number analyzed (Participants) | 210
Number analyzed (limbs) | 275
Percentage of limbs | 94.0 (1.3)

12. Primary Outcome: Percentage of Limbs Without Reflux in the Treated Vein Segment
Description: as for outcome 7
Time Frame: 5 years
Population: 279 limbs were evaluated at the 5Y timepoint
Measure: Mean (Standard Error); unit: Percentage of limbs
Units Other Than Participants: limbs
Arm/Group | ClosureFAST® - Endovascular Radiofrequency Great Saphenous Vei
Number analyzed (Participants) | 221
Number analyzed (limbs) | 279
Percentage of limbs | 93.7 (1.3)

13. Secondary Outcome: CEAP (Clinical, Etiologic, Anatomic, and Pathophysiologic) Classification
Description: Status of clinical signs and symptoms of lower limb venous disease as measured by CEAP Classification at baseline. The CEAP clinical Categories are as follows where C1 is of the least clinical concern and C6 is the worst stage; C1- Reticular and spider veins C2- Varicose veins C3- Varicose veins and leg swelling C4- Varicose veins and evidence of venous stasis skin changes C5- Varicose veins and a healed venous stasis ulceration C6- Varicose veins and an open venous ulceration
  Reference: Kistner RL, Eklof B, Masuda EM. Diagnosis of chronic venous disease of the lower extremities: The "CEAP" classification. Mayo Clinic Proc 1996;71:338-45.
Time Frame: Baseline
Measure: Count of Units; unit: limbs
Units Other Than Participants: limbs
Arm/Group | ClosureFAST® - Endovascular Radiofrequency Great Saphenous Vei
Number analyzed (Participants) | 326
Number analyzed (limbs) | 395
limbs
  C0 | 1
  C1 | 5
  C2 | 213
  C3 | 110
  C4 | 60
  C5 | 4
  C6 | 2

14. Secondary Outcome: CEAP Classification
Description: Status of clinical signs and symptoms of lower limb venous disease as measured by CEAP Classification at follow-up where C1 is the best and C6 is the worst in terms of clinical status.
Time Frame: 1 Week
Measure: Count of Units; unit: limbs
Units Other Than Participants: limbs
Arm/Group | ClosureFAST® - Endovascular Radiofrequency Great Saphenous Vei
Number analyzed (Participants) | 325
Number analyzed (limbs) | 395
limbs
  C0 | 55
  C1 | 180
  C2 | 92
  C3 | 27
  C4 | 36
  C5 | 3
  C6 | 2

15. Secondary Outcome: CEAP Classification
Description: as for outcome 14
Time Frame: 3 months
Population: Only 302 subjects (371 limbs) completed the 3 Month follow-up visit to provide data to this outcome measure.
Measure: Count of Units; unit: limbs
Units Other Than Participants: limbs
Arm/Group | ClosureFAST® - Endovascular Radiofrequency Great Saphenous Vei
Number analyzed (Participants) | 302
Number analyzed (limbs) | 371
limbs
  C0 | 67
  C1 | 173
  C2 | 84
  C3 | 10
  C4 | 35
  C5 | 1
  C6 | 1

16. Secondary Outcome: CEAP Classification
Description: as for outcome 14
Time Frame: 12 months
Population: Only 280 subjects (350 limbs) completed the 12 Month follow-up visit to provide data to this outcome measure.
Measure: Count of Units; unit: limbs
Units Other Than Participants: limbs
Arm/Group | ClosureFAST® - Endovascular Radiofrequency Great Saphenous Vei
Number analyzed (Participants) | 280
Number analyzed (limbs) | 350
limbs
  C0 | 62
  C1 | 194
  C2 | 61
  C3 | 6
  C4 | 24
  C5 | 2
  C6 | 1

17. Secondary Outcome: CEAP Classification
Description: as for outcome 14
Time Frame: 5 years
Population: Only 221 subjects (279 limbs) completed the 5 Year follow-up visit to provide data to this outcome measure.
Measure: Count of Units; unit: limbs
Units Other Than Participants: limbs
Arm/Group | ClosureFAST® - Endovascular Radiofrequency Great Saphenous Vei
Number analyzed (Participants) | 221
Number analyzed (limbs) | 279
limbs
  C0 | 22
  C1 | 116
  C2 | 101
  C3 | 26
  C4 | 12
  C5 | 2
  C6 | 0

18. Secondary Outcome: Change in Venous Clinical Severity Score (VCSS) From Baseline to 5Y Follow-up
Description: Status of clinical signs and symptoms of lower limb venous disease evaluated using standardized scales and subject responses to post-procedure standardized questions - VCSS Status from Baseline to 5 years. VCSS assesses 10 factors of venous disease whereby each factor is graded on a severity scale of 0-3 (least to worst). The higher the VCSS score the most severe the clinical signs and symptoms of venous disease are in a patient. VCSS improvement over time is presented by a decrease in VCSS total score (maximum score = 30; minimum score = 0).
  Reference: Rutherford RB, Padberg FT Jr, Comerota AJ, Kistner RL, Meissner MH, Moneta GL. Venous severity scoring: An adjunct to venous outcome assessment. J Vasc Surg 2000;31:1307-12.
Time Frame: Baseline thru 5 years
Measure: Mean (Standard Deviation); unit: VCSS Score
Units Other Than Participants: limbs
Arm/Group | ClosureFAST® - Endovascular Radiofrequency Great Saphenous Vei
Number analyzed (Participants) | 326
Number analyzed (limbs) | 396
VCSS Score
  Baseline | 4.4 (2.5)
  1 week | 4.1 (1.7)
  3 months | 1.3 (1.8)
  6 months | 1.0 (1.5)
  12 months | 0.9 (1.6)
  2 years | 0.9 (1.5)
  3 years | 1.1 (1.5)
  4 years | 1.0 (1.4)
  5 years | 1.5 (1.8)

19. Secondary Outcome: Visual Analog Pain Scale (VAS)
Description: Status of clinical signs and symptoms of lower limb venous disease evaluated using standardized scales and subject responses to post-procedure standardized questions - VAS for pain scored from 0-10 with 10 being worst possible pain
Time Frame: 5 years
Measure: Mean (Standard Deviation); unit: units on a scale (0-10)
Units Other Than Participants: limbs
Arm/Group | ClosureFAST® - Endovascular Radiofrequency Great Saphenous Vei
Number analyzed (Participants) | 326
Number analyzed (limbs) | 395
units on a scale (0-10)
  1 week | 1.2 (1.9)
  3 months | 0.4 (1.2)
  6 months | 0.2 (0.8)
  12 months | 0.2 (1.1)
  2 years | 0.2 (0.7)
  3 years | 0.2 (1.0)
  4 years | 0.1 (1.0)
  5 years | 0.2 (1.1)

20. Secondary Outcome: Presence of Complications From Greater Saphenous Vein (GSV) Intervention
Description: Number of limbs that presented with the listed complications and side effects resulting from the GSV intervention.
Time Frame: 1 Week
Measure: Count of Units; unit: limbs
Units Other Than Participants: limbs
Arm/Group | ClosureFAST® - Endovascular Radiofrequency Great Saphenous Vei
Number analyzed (Participants) | 326
Number analyzed (limbs) | 395
limbs
  Ecchymosis | 23
  Erythema | 5
  Hematoma | 4
  Infection | 0
  Pain | 7
  Paresthesia | 6
  Phlebitis | 5
  Skin Pigmentation | 0
  Thermal Skin Injury | 0
  Thrombus Extension / DVT | 6

21. Secondary Outcome: Presence of Complications From GSV Intervention
Description: Number of limbs that presented with the listed complications and side effects resulting from the GSV intervention.
Time Frame: 3 Months
Measure: Count of Units; unit: limbs
Units Other Than Participants: limbs
Arm/Group | ClosureFAST® - Endovascular Radiofrequency Great Saphenous Vei
Number analyzed (Participants) | 326
Number analyzed (limbs) | 371
limbs
  Ecchymosis | 0
  Erythema | 0
  Hematoma | 1
  Infection | 0
  Pain | 0
  Paresthesia | 9
  Phlebitis | 1
  Skin Pigmentation | 4
  Thermal Skin Injury | 0
  Thrombus Extension / DVT | 3

22. Secondary Outcome: Presence of Complications From GSV Intervention
Description: Number of limbs that presented with the listed complications and side effects resulting from the GSV intervention.
Time Frame: 12 months
Measure: Count of Units; unit: limbs
Units Other Than Participants: limbs
Arm/Group | ClosureFAST® - Endovascular Radiofrequency Great Saphenous Vei
Number analyzed (Participants) | 326
Number analyzed (limbs) | 350
limbs
  Ecchymosis | 0
  Erythema | 0
  Hematoma | 0
  Infection | 0
  Pain | 2
  Paresthesia | 1
  Phlebitis | 0
  Skin Pigmentation | 3
  Thermal Skin Injury | 0
  Thrombus Extension / DVT | 1

23. Secondary Outcome: Presence of Complications From GSV Intervention
Description: Number of limbs that presented with the listed complications and side effects resulting from the GSV intervention.
Time Frame: 5 years
Measure: Count of Units; unit: limbs
Units Other Than Participants: limbs
Arm/Group | ClosureFAST® - Endovascular Radiofrequency Great Saphenous Vei
Number analyzed (Participants) | 326
Number analyzed (limbs) | 279
limbs
  Ecchymosis | 0
  Erythema | 0
  Hematoma | 0
  Infection | 0
  Pain | 1
  Paresthesia | 2
  Phlebitis | 0
  Skin Pigmentation | 1
  Thermal Skin Injury | 0
  Thrombus Extension / DVT | 0

ADVERSE EVENTS:
Time Frame: 5 years
Description: SAEs were collected through study closure at 5 years. An SAE was defined as any AE that led to death, to a serious deterioration in the health of a subject that resulted in a life-threatening injury, a permanent impairment of a body structure/body function, hospitalization or prolongation of existing hospitalization, in a medical or surgical intervention to prevent permanent impairment of body structures or a body function; or led to fetal distress, fetal death, or a congenital birth defect.
Arm/Group | ClosureFAST® - Endovascular Radiofrequency Great Saphenous Vei
All-Cause Mortality (participants affected / at risk) | 2/326
Serious Adverse Events (participants affected / at risk) | 10/326
Other Adverse Events (participants affected / at risk) | 0/326
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ClosureFAST® - Endovascular Radiofrequency Great Saphenous Vei (N=326)
GI Bleed (Gastrointestinal disorders) | 1 (1) — Unrelated event, Fatal GI Bleed
Thrombus extensions (Vascular disorders) | 6 (6) — Thrombus extensions into the Common Femoral vein (CFV)
Pulmonary Emboli (PE) (Vascular disorders) | 1 (1) — Pulmonary Emboli (PE)
Death (Unknown Cause) (General disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less